CLINICAL TRIAL: NCT05624931
Title: Reducing Psychological Barriers to PrEP Persistence Among Pregnant and Postpartum Women in Cape Town, South Africa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: University of Cape Town (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6783E; K23MH131438 (NIH)
Record Dates: First submitted 2022-10-31; First posted 2022-11-22 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Depression; Posttraumatic Stress Disorder; Pregnancy Related; Medication Adherence
Keywords: HIV, pregnancy, PrEP
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Aims 1 and 2 will assess a single group of pregnant women. In Aim 3, a randomized control trial will include an intervention group and control group that are running in parallel.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Condition: Brief CBT-Based Intervention (Experimental): This group (n=30) will be guided through an adaptation of Life Steps, a single-session, cognitive behavioral therapy (CBT)-based medication adherence intervention that has been used to increase PrEP adherence. Participants will also receive four additional intervention sessions.
  Interventions: Behavioral: Brief CBT-Based Intervention
- Control Condition: Enhanced Treatment as Usual (Active Comparator): Participants randomized to the control condition (n= 30) will receive enhanced treated as usual.
  Interventions: Other: Enhanced Treatment as Usual

INTERVENTIONS:
Behavioral: Brief CBT-Based Intervention — Aims 1 (n=30) and 2 (n=18) will inform the Aim 3 intervention. We anticipate that the intervention will be comprised of four treatment sessions. These sessions will likely target two pathways to PrEP adherence and persistence: (1) decreased withdrawal and avoidance and (2) behavioral skill building to increase self-care/health behaviors. To decrease withdrawal and avoidance, we will likely include CBT-based exercises that improve distress tolerance and coping. To help participants build new behavioral skills, we will likely incorporate behavioral activation and problem-solving. Behavioral activation is a CBT strategy that promotes scheduling activities that align with an individual's values, which will also break maladaptive patterns of withdrawal and avoidance. Problem-solving is an empirically-supported treatment for depression; training patients to problem-solve adaptively will help them "approach" PrEP use by navigating barriers.
  Arms: Treatment Condition: Brief CBT-Based Intervention
Other: Enhanced Treatment as Usual — This is the control intervention. Participants will receive antenatal care as usual, which is monthly visits to the MOU, information about using PrEP during pregnancy (information sheet or pamphlet), and a psychological services referral.
  Arms: Control Condition: Enhanced Treatment as Usual

SUMMARY:
Pregnant women in South Africa (SA) are at high risk of HIV acquisition. Pre-exposure prophylaxis (PrEP) use during pregnancy is both safe and effective in preventing HIV. However, posttraumatic stress (associated with intimate partner violence and/or other traumas) and depression negatively impact PrEP adherence among women in SA. Addressing posttraumatic stress and depression will likely improve PrEP adherence and persistence (i.e., sustained PrEP adherence over time) during pregnancy and breastfeeding, which are periods of dramatically increased HIV risk. The overarching goal of this proposal is to develop and test the feasibility and acceptability of a cognitive behavioral intervention that targets common underlying factors of posttraumatic stress and depression to improve PrEP adherence and persistence during pregnancy and the postpartum transition. The specific aims of the project are to (1) explore the mechanisms by which posttraumatic stress and depression impact PrEP adherence and persistence during pregnancy via qualitative interviews; (2) develop a brief PrEP adherence and persistence intervention (~4 sessions) that reduces the negative impact of psychological mechanisms common to posttraumatic stress and depression on PrEP use, and builds behavioral skills to improve self-care; and (3) evaluate the feasibility, acceptability, and signals of preliminary efficacy of the intervention, which will be integrated into antenatal care, in a pilot randomized controlled trial. All data will be collected in the Midwife Obstetrics Unit (MOU) in Gugulethu, a peri-urban settlement and former township community outside of Cape Town, SA.

ELIGIBILITY:
Inclusion Criteria:

* For participants across all three aims are:

  * Female sex
  * Aged 15+
  * Pregnant and presenting antenatal care at the Gugulethu MOU
  * HIV-negative
  * Recent PrEP initiation (<1 month ago) or PrEP adherence challenges, either documented (>2 weeks late to pick up PrEP refill) or self-reported
  * Moderate to severe symptoms of posttraumatic stress and/or depression (defined as a score of ≥31 on PTSD Checklist for DSM-5 (PCL-5) and/or a score of ≥13 on the Edinburgh Postnatal Depression Scale (EPDS). Cutoff scores may be adjusted by 3-5 points to facilitate recruitment.

Exclusion Criteria:

* There are no exclusion criteria with respect to parity or gravidity.

  * Participants who are unable to provide informed consent or assent in English or Xhosa
  * Have a significant psychiatric illness (e.g., active psychotic disorder or untreated bipolar disorder) that could interfere with participation will be excluded. Positive symptoms of active psychosis or mania will be assessed by the research assistants. They will be trained to identify delusions, hallucinations, disorganized or pressured speech, flight of ideas, and grandiosity as they speak to potential participants.
  * Potential participants will also be asked if they have any health conditions that make it difficult for them to travel to the clinic.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention | This will be assessed at 2 months post-baseline
  Feasibility will be assessed by (1) interventionist fidelity to the protocol, (2) treatment session attendance, and (3) participant retention at 3-months postpartum (T3). Feasibility will be demonstrated if at least (1) 80% of the reviewed sessions addressed 90% of the key session components, (2) 75% of the participants (at least 23 of 30) attended at least two of the four treatment sessions; and (3) 60% of the participants (at least 18 of 30) completed the three-month postpartum assessment (T3). To measure fidelity, we will review 20% of the session audio-recordings randomly selected from each of the four sessions and determine whether key session components were addressed.
Acceptability | This will be assessed at 2 months post-baseline
  Acceptability will be assessed (1) in the qualitative exit interviews and (2) with the brief acceptability questionnaire completed after each intervention session. Acceptability data from the qualitative exit interviews will be described, and the intervention will be deemed acceptable if at least 75% of the participants rate three or more of the items on the acceptability questionnaires with "high satisfaction" (4 or 5 on the Likert-style scale).

SECONDARY OUTCOMES:
PrEP Adherence | This will be assessed at 2 months post-baseline and at 3 months postpartum
  PrEP adherence during the previous week will be assessed at the end of the intervention/2 months post-baseline (T2) and at 3-months postpartum (T3) via an adapted version of the Wilson three-item self-report adherence scale, which includes (1) number of missed doses, (2) the percentage of time that PrEP was taken as prescribed, and (3) a rating of one's ability to take PrEP.
PrEP Persistence | This will be assessed at 2 months post-baseline and at 3 months postpartum
  PrEP persistence at T2 and T3 will be determined via dried blood spot (DBS) testing and defined as tenofovir- diphosphate (TVF-DP) concentrations of at least 650 fmol/punch for pregnant women and 1050 fmol/punch for postpartum women, which are indicative of 7 doses per week over a period of up to eight weeks.
Posttraumatic Stress Disorder (PTSD) | This will be assessed at 2 months post-baseline and at 3 months postpartum
  Changes in PTSD symptom severity from baseline will be measured using the PTSD Checklist for DSM-5 (PCL-5). A cutoff score of ≥31 will be used to determine moderate or severe PTSD symptoms.
Depression | This will be assessed at 2 months post-baseline and at 3 months postpartum
  Changes in depression from baseline will be measured using the Edinburgh Postnatal Depression Scales. A cutoff score of ≥13 will be used to determine moderate or severe depression symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Stanton, PhD, Principal Investigator — Boston University
Locations (2):
- Boston University, Boston, Massachusetts, United States
- Gugulethu Midwife Obstetric Unit (MOU), Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No